CLINICAL TRIAL: NCT03511443
Title: Evaluation of the Performance of a Highly-sensitive Rapid Diagnostic Test (RDT) Versus Conventional RDT, Compared With PCR as the Gold Standard, in Reactive Case Detection of Malaria Infections in Rakhine State, Myanmar
Brief Title: Evaluation of the Performance of a hsRDT Versus cRDT in Reactive Case Detection of Malaria Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Research Co, LLC (Industry)
Collaborators: Duke University (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Department of Medical Research, Lower Myanmar (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00076579; Pro00089928 (Other: Duke University)
Record Dates: First submitted 2018-03-19; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Malaria Diagnosis; Malaria,Falciparum
Keywords: hsRDT; usRDT; Reactive Case Detection (RCD); High risk for malaria
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: If P.f malaria case were detected, the responsible malaria worker or basic health staff will inform to survey team and blood samples for cRDT, hsRDT, Dried Blood Spot for PCR will be collected from index case and contacts (nearby 10-household members and peers). Then the results of cRDT and hsRDT will be confirmed by PCR for evaluating their performance. Then the applicability of hsRDT to detect low parasitaemia for enhancing malaria elimination activities will be evaluated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic performance of hsRDT (Other): Comparing diagnostic power of two diagnostics
  Interventions: Diagnostic Test: hsRDT

INTERVENTIONS:
Diagnostic Test: hsRDT — Testing highly sensitive RDT detection for low parasitemia
  Other Names: Highly sensitive RDT is also used as ultrasensitive RDT

SUMMARY:
A systematic review assessing the role, appropriateness and benefits of the active case detection strategy, both proactive and reactive, in low malaria transmission settings. A common indication is that more studies should be carried out to optimize the ACD strategy to the local context, or to provide evidence for the adoption of improved methods. One possible improved method is the use of more accurate diagnostic tools, such as the hsRDT proposed in this study, with an increased capacity to detect lower levels of parasitemia. It can provide a timely and relevant contribution for their development of national Standard Operating Procedures for a screening tool in the reactive case detection strategy.

DETAILED DESCRIPTION:
The study is conducted in the areas under Sakhanmaw Rural Health Center, Ann Township in Southern Rakhine State, Myanmar.

General objective was to evaluate the performance of the new highly-sensitive rapid diagnostic test (RDT) developed by SD Bioline versus conventional RDT, compared with PCR as the gold standard, in reactive case detection of malaria infections in Rakhine State, Myanmar.

Specific objectives

* To evaluate the prevalence of malaria identified by the new hsRDT in comparison with that by cRDT and PCR
* To assess the diagnostic performance characteristics of hsRDT versus cRDT, using PCR as gold standard, in the detection of P.falciparum infections
* To evaluate correlation of detection capability between cRDT and hsRDT
* To identify risk factors associated with malaria infection, including but not limited to, socio-demographic factors and travel history related with malaria index cases

This is a prospective community-based single-center reactive case detection (RCD) study to assess the performance of hsRDT versus cRDT in identifying individuals with malaria infection ("Secondary case") in a population living and/or working in a close physical proximity to an "index case." All cases parasitologically confirmed by conventional RDT will be promptly notified to the study team and interviewed with a standardized case investigation form at their home, possibly within 3 days. All members of the primary case household and those of the nearest 10 households, aged 5 years and above, will be invited to participate in the study. A blood spot will be collected for subsequent PCR analysis. At least 50 index cases are targeted for investigation and reactive case detection and an estimated number of 1,980 persons will be involved in the study.

It is expected that this study will be an important input for the national malaria control program in Myanmar as they develop the strategies to conduct reactive case detection.

A suitable statistical software, e.g. STATA will be used to analyze the data resulting from the participant interviews and 3 parasitological tests. Logistic regression models will be developed to examine factors significantly associated with malaria infections.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 5 years old
* Resident of the villages, or temporary visitors, or co-workers or co-travelers of index case
* Willingness to participate in the study evident by informed consent

Exclusion Criteria:

* Presence of severe clinical illness including severe malaria
* Non-resident index cases
* Refusal to participate in the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1980 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-06-28 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malaria infections identified by the new hsRDT | PCR diagnosis of samples will occur after 10 months of data collection.
  Outcomes measured by malaria test positivity rate by cRDT, hsRDT and PCR, respectively

SECONDARY OUTCOMES:
Diagnostic performance characteristics of hsRDT versus cRDT using PCR as gold standard, in the detection of P.falciparum infections | Outcomes will be analyzed after 10 months of data collection
  Outcomes measured between hsRDT and cRDT
Correlation of detection capability between cRDT and hsRDT | PCR results will be analyzed during month 10
  Outcomes measured by correlation of test positivity rates
Risk factors associated with malaria infection cases | Outcome will be measured/analyzed in month 10, after PCR results are released
  Outcomes will be measured by relative risk of malaria in association with different risk factors identified

CONTACTS AND LOCATIONS:
Overall Officials: Saw Lwin, MD, Study Chair — University Research Co, LLC; Feliciano Monti, MD, Study Chair — US Embassy, Yangon
Locations (1):
- University Research Co., LLC (URC), Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen I, Clarke SE, Gosling R, Hamainza B, Killeen G, Magill A, O'Meara W, Price RN, Riley EM. "Asymptomatic" Malaria: A Chronic and Debilitating Infection That Should Be Treated. PLoS Med. 2016 Jan 19;13(1):e1001942. doi: 10.1371/journal.pmed.1001942. eCollection 2016 Jan. PMID 26783752
- [Background] malERA Consultative Group on Health Systems and Operational Research. A research agenda for malaria eradication: health systems and operational research. PLoS Med. 2011 Jan 25;8(1):e1000397. doi: 10.1371/journal.pmed.1000397. PMID 21311588
- [Background] Adams M, Joshi SN, Mbambo G, Mu AZ, Roemmich SM, Shrestha B, Strauss KA, Johnson NE, Oo KZ, Hlaing TM, Han ZY, Han KT, Thura S, Richards AK, Huang F, Nyunt MM, Plowe CV. An ultrasensitive reverse transcription polymerase chain reaction assay to detect asymptomatic low-density Plasmodium falciparum and Plasmodium vivax infections in small volume blood samples. Malar J. 2015 Dec 23;14:520. doi: 10.1186/s12936-015-1038-z. PMID 26701778
- [Background] Cheng Z, Wang D, Tian X, Sun Y, Sun X, Xiao N, Zheng Z. Capture and Ligation Probe-PCR (CLIP-PCR) for Molecular Screening, with Application to Active Malaria Surveillance for Elimination. Clin Chem. 2015 Jun;61(6):821-8. doi: 10.1373/clinchem.2014.237115. Epub 2015 May 11. PMID 25964304
- [Background] Okell LC, Ghani AC, Lyons E, Drakeley CJ. Submicroscopic infection in Plasmodium falciparum-endemic populations: a systematic review and meta-analysis. J Infect Dis. 2009 Nov 15;200(10):1509-17. doi: 10.1086/644781. PMID 19848588
- [Background] Imwong M, Hanchana S, Malleret B, Renia L, Day NP, Dondorp A, Nosten F, Snounou G, White NJ. High-throughput ultrasensitive molecular techniques for quantifying low-density malaria parasitemias. J Clin Microbiol. 2014 Sep;52(9):3303-9. doi: 10.1128/JCM.01057-14. Epub 2014 Jul 2. PMID 24989601
- [Background] Imwong M, Nguyen TN, Tripura R, Peto TJ, Lee SJ, Lwin KM, Suangkanarat P, Jeeyapant A, Vihokhern B, Wongsaen K, Van Hue D, Dong le T, Nguyen TU, Lubell Y, von Seidlein L, Dhorda M, Promnarate C, Snounou G, Malleret B, Renia L, Keereecharoen L, Singhasivanon P, Sirithiranont P, Chalk J, Nguon C, Hien TT, Day N, White NJ, Dondorp A, Nosten F. The epidemiology of subclinical malaria infections in South-East Asia: findings from cross-sectional surveys in Thailand-Myanmar border areas, Cambodia, and Vietnam. Malar J. 2015 Sep 30;14:381. doi: 10.1186/s12936-015-0906-x. PMID 26424000
- [Background] Searle KM, Shields T, Hamapumbu H, Kobayashi T, Mharakurwa S, Thuma PE, Smith DL, Glass G, Moss WJ. Efficiency of household reactive case detection for malaria in rural Southern Zambia: simulations based on cross-sectional surveys from two epidemiological settings. PLoS One. 2013 Aug 6;8(8):e70972. doi: 10.1371/journal.pone.0070972. Print 2013. PMID 23940677
- [Background] van Eijk AM, Ramanathapuram L, Sutton PL, Kanagaraj D, Sri Lakshmi Priya G, Ravishankaran S, Asokan A, Tandel N, Patel A, Desai N, Singh R, Sullivan SA, Carlton JM, Srivastava HC, Eapen A. What is the value of reactive case detection in malaria control? A case-study in India and a systematic review. Malar J. 2016 Feb 6;15:67. doi: 10.1186/s12936-016-1120-1. PMID 26852118
- [Background] Hustedt J, Canavati SE, Rang C, Ashton RA, Khim N, Berne L, Kim S, Sovannaroth S, Ly P, Menard D, Cox J, Meek S, Roca-Feltrer A. Reactive case-detection of malaria in Pailin Province, Western Cambodia: lessons from a year-long evaluation in a pre-elimination setting. Malar J. 2016 Mar 1;15:132. doi: 10.1186/s12936-016-1191-z. PMID 26931488

DOCUMENTS (2):
  • Informed Consent Form (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03511443/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT03511443/Prot_SAP_001.pdf